CLINICAL TRIAL: NCT04502979
Title: Enhancing Caregiver-Infant Communication to Prevent Obesity
Brief Title: Learning to Love Mealtime Together
Acronym: LiTTLe Me
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 15-2437; R21HD082707 (NIH)
Record Dates: First submitted 2020-07-29; First posted 2020-08-06 (Actual); Results first posted 2020-09-11 (Actual); Last update posted 2020-09-11 (Actual); Status verified 2020-08

CONDITIONS: Infant Obesity; Parenting; Feeding Behavior
Keywords: Infant Obesity; Parenting; Feeding Behavior; Responsive Feeding
MeSH Terms: conditions — Pediatric Obesity; Feeding Behavior

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Responsive Feeding (Experimental): Intervention families will receive approximately 4 hours of ASL and development specific content related to language and feeding during home visits and phone calls. The initial in-home session with families will focus on teaching ASL signs indicative of hunger, thirst, and satiety. A video and placemat of mealtime signs will be left with families at the completion of the first visit. The remaining sessions, in-home over the next 3 months and by phone monthly thereafter for 6 months total, will focus on reinforcing ASL signing in addition to focused education on particular aspects of language development (receptive language preceding expressive language and increasing intentional communication), feeding development (such as hunger and fullness cues, fear of new foods, the importance of repeated food exposures, variations in intake from meal-to-meal, and the propensity to reject bitter tastes [many vegetables]55], and appropriate portion sizes and variety for healthy growth.
  Interventions: Behavioral: Responsive Feeding Training
- Routine Care (No Intervention): No intervention is provided to the families in this group; however, portions of the intervention lessons will be made available after completion of data collection.

INTERVENTIONS:
Behavioral: Responsive Feeding Training — Families will receive 4 monthly 1-hour sessions: (1) Signing with infants; (2) infant communication and responsive feeding; (3) nutrition, portion sizes, and neophobia; and, (4) infant intentionality.
  Arms: Responsive Feeding

SUMMARY:
Infancy is an important target period for obesity prevention because once obese as an infant, the relative risk of remaining obese appears to rise with increasing age at great cost to both individuals and society. The ability to self-regulate energy intake (eating when hungry and stopping when full) is vital to obesity prevention and it is thought that this ability can be derailed by a chronic mismatch between parental feeding behavior and the infant's state (feeding in the absence of hunger and/or feeding beyond fullness). The study will test a novel intervention to help parents and pre-verbal infants better understand one another during feeding and it will offer new insight into how self-regulation of energy intake develops during infancy.

DETAILED DESCRIPTION:
Once obese as an infant, the relative risk of remaining obese appears to rise with increasing age. Thus, the early years of life have been posited as an important target period for obesity prevention. Widely viewed as a response to genetic, interpersonal, and environmental factors, obesity fundamentally reflects an imbalance between energy intake and expenditure. Self-regulation of energy intake aligned with physiologic need is essential to this balance. The process(es) by which infants begin to disassociate eating behavior from physiologic need is unclear, thus it is crucial to better understand predictors of individual differences in self-regulation of energy intake. It is well established that autonomic regulation may support infant behavioral regulation, suggesting that autonomic function may be a critical area to consider here. Moreover, self-regulation is strongly influenced by dyadic interaction quality during infancy, and findings reveal that more responsive interactions are associated with more effective autonomic regulation. A chronic mismatch between a caregiver's feeding behavior and the infant's state (feeding in the absence of hunger and/or feeding beyond fullness), is thought to contribute to obesity by undermining the infant's capacity to self-regulate intake; the current proposal will be the first to examine the effects on autonomic regulation. The investigators propose an intervention to enrich the capacity of mother-infant dyads to perform their respective interactive tasks. The investigators plan to teach mothers American Sign Language (ASL) signs indicative of hunger, thirst, and satiety, which they will in turn teach their preverbal infant. This training in ASL will be augmented with targeted information for mothers about infants' capacities to self-regulate energy intake in response to hunger and satiety and communicate those states with intention. Mothers also will be taught about expected development of infants' eating behaviors and nutritional requirements to support healthy growth.

Using a two-group randomized repeated measures design, this study aims to 1) evaluate the feasibility and acceptability of the intervention and study methods, including recruitment, enrollment, and data collection (self-report, anthropometrics, video observations, and respiratory sinus arrhythmia [RSA]) for infants and their mothers; 2) evaluate the initial impact of the intervention on observed feeding interactions, reported infant feeding behaviors and maternal feeding behaviors/beliefs, and infant nutritional intake and growth; and, 3) explore preliminary data on concordance between dyadic feeding interactions and autonomic regulation in both mothers and infants (RSA). In addition to a variety of self-report and anthropometric measures, this study will use integrated behavioral (video) and physiologic (RSA) measures to better understand feeding dynamics and their relationship with obesity risk. Understanding these processes is essential for developing appropriate preventions, or interventions, that will help reduce the prevalence of early childhood obesity and its extension into later childhood and beyond.

Study Phases:

Screening: screening for eligibility and obtaining consent

Study Treatment: study intervention/experimental treatment from baseline visit ([Time 1 (T1)]: age 4-9-months) monthly until 3-months post-baseline ([Time 2 (T2)]: age 7-12-months)

Follow-up: 6-months post-baseline ([Time 3 (T3)]: age 10-15-months)

ELIGIBILITY:
Inclusion Criteria:

Parent Inclusion:

* Must be able to read, understand, and speak English or Spanish and be willing to be randomized and participate in data collection.
* Those who are randomized into the experimental group must also be willing to learn ASL specific to communication of hunger, thirst, and fullness.

Infant Inclusion:

* Aged at least 3 months at the time of recruitment

Exclusion Criteria:

Parent Exclusion:

* > 50 years of age

Infant Exclusion:

* Aged more than 9 months at the time of recruitment
* born more than 6 weeks earlier than their estimated due date,
* have any developmental delays or disabilities that make it difficult for them to eat, drink, or communicate,
* attend regular daycare,
* will be younger than 4 months or older than 9 months at the time of the first ASL training.

Ages: 3 Months to 9 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 71 (Actual)
Dates: Start 2017-09-26 (Actual); Primary Completion 2019-04-11 (Actual); Study Completion 2019-04-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Hodges, PhD, FNP-BC, FAAN, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with The University of North Carolina at Chapel Hill (UNC).
Time Frame: 9 to 36 months following publication
Access Criteria: The investigator proposing to use the data has approval from an IRB, IEC, or REB, as applicable, and an executed data use/sharing agreement.

RESULTS

PARTICIPANT FLOW:
Groups:
- Responsive Feeding: Intervention families will receive approximately 4 hours of American Sign Language (ASL) and development-specific content related to language and feeding during home visits and phone calls. The initial in-home session with families focused on teaching ASL signs indicative of hunger, thirst, and satiety. A video and placemat of mealtime signs are left with families at the end of the first visit. The remaining sessions, in-home over the next 3 months and by phone monthly thereafter for 6 months total, will focus on reinforcing ASL signing in addition to focused education on particular aspects of language development (receptive language preceding expressive language and increasing intentional communication), feeding development (such as hunger and fullness cues, fear of new foods, the importance of repeated food exposures, variations in intake from meal-to-meal, and the propensity to reject bitter tastes [many vegetables], and appropriate portion sizes and variety for healthy growth.
Period: Overall Study
Arm/Group | Responsive Feeding | Routine Care
Started | 37 | 34
Completed | 34 | 30
Not Completed | 3 | 4
Not completed — Lost to Follow-up | 1 | 3
Not completed — Withdrawal by Subject | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Responsive Feeding: Intervention families will receive approximately 4 hours of ASL and development specific content related to language and feeding during home visits and phone calls. The initial in-home session with families will focus on teaching ASL signs indicative of hunger, thirst, and satiety. A video and placemat of mealtime signs will be left with families at the completion of the first visit. The remaining sessions, in-home over the next 3 months and by phone monthly thereafter for 6 months total, will focus on reinforcing ASL signing in addition to focused education on particular aspects of language development (receptive language preceding expressive language and increasing intentional communication), feeding development (such as hunger and fullness cues, fear of new foods, the importance of repeated food exposures, variations in intake from meal-to-meal, and the propensity to reject bitter tastes [many vegetables], and appropriate portion sizes and variety for healthy growth.
- Total: Total of all reporting groups
Arm/Group | Responsive Feeding | Routine Care | Total
Number analyzed (Participants) | 37 | 34 | 71
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 37 | 34 | 71
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: months] | 6.86 (1.57) | 7.29 (1.64) | 7.07 (1.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 19 | 34
  Male | 22 | 15 | 37
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 3 | 8
  Not Hispanic or Latino | 32 | 31 | 63
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 9 | 14
  White | 23 | 20 | 43
  More than one race | 6 | 4 | 10
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 37 | 34 | 71

OUTCOME MEASURES:

1. Primary Outcome: Infant Weight-for-Length Z Scores
Description: The infant's length and weight (in clean dry diaper only) will be measured in triplicate, using a calibrated length board and digital scale. The mean of the three length measurements (cm) and the mean of the three weight measurements (kg) will be combined to report a sex-specific weight-for-length z score. Weight-for-Length Z scores are measures of relative weight adjusted for child length and sex. The Z-score indicates the number of standard deviations away from a reference population in the same age range and with the same sex. A Z-score of 0 is equal to 50th percentile (median). Negative numbers indicate values lower than the median and positive numbers indicate values higher than the median.
Time Frame: 6 Months Post-Baseline (T3)
Population: Measurement error resulted in improbable length data (length recorded as shorter than length at prior visit when infant was younger) for 10 infants total (Responsive Feeding n = 6; Routine Care n = 4). Data for these 10 infants were excluded from analysis at T3.
Measure: Mean (Standard Error); unit: z-score
Arm/Group | Responsive Feeding | Routine Care
Number analyzed (Participants) | 28 | 26
z-score | 0.43 (0.15) | 0.12 (0.15)
Statistical Analysis 1: Comparison: Responsive Feeding vs Routine Care; Test type: Superiority; p = 0.07, Mixed Models Analysis — One-sided p-value for directional hypothesis. The threshold for statistical significance is p < 0.05; Mean Difference (Net) = 0.31, 95% CI 2-sided [-0.11 to 0.73], Standard Error of Mean 0.21

2. Secondary Outcome: Mean Infant Caloric Intake Compared to Estimated Energy Requirements
Description: Group mean of Kcal difference between dietary recall (mean of total Kcal from 2-day 24-hour recalls calculated in the Nutrition Data System for Research (NDS-R)) and age-and-sex-specific estimated energy requirements. Lower values represent greater precision of intake.
Time Frame: 6 Months Post-Baseline (T3)
Population: All data reported were included (missing for 13 infants).
Measure: Mean (Standard Error); unit: Kcal
Arm/Group | Responsive Feeding | Routine Care
Number analyzed (Participants) | 32 | 26
Kcal | 120.90 (43.37) | 242.06 (48.73)
Statistical Analysis 1: Comparison: Responsive Feeding vs Routine Care; Test type: Superiority; p = 0.04, Mixed Models Analysis — One-sided p-value for directional hypothesis. The threshold for statistical significance is p < 0.05; Mean Difference (Net) = -121.16, 95% CI 2-sided [-252.73 to 10.41], Standard Error of Mean 65.73

ADVERSE EVENTS:
Time Frame: From Baseline through Study Completion, an approximate total of 6 months
Arm/Group | Responsive Feeding | Routine Care
All-Cause Mortality (participants affected / at risk) | 0/37 | 0/34
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/34
Other Adverse Events (participants affected / at risk) | 0/37 | 0/34

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-01): https://cdn.clinicaltrials.gov/large-docs/79/NCT04502979/Prot_SAP_000.pdf